## 1. TITLE PAGE

| <b>Protocol Title:</b> | Clinical Pilot Study to Provide Research Data for TONOREF |
|---|---|
| | III Tested to ANSI Z80.10-2014 |
| <b>Protocol Number:</b> | NIDEK-TONOREF-PILOT-0002 |
| <b>Product Name:</b> | Auto ref/kerato/tono/pachymeter TONOREF III |
| <b>Proposed Indications</b> | The auto ref/kerato/tono/pachymeter TONOREF III is a |
| for use: | medical device which measures objective refractive errors, |
| | corneal curvature radius, intraocular pressure and corneal |
| | thickness of the patient's eye. |
| Site/Investigators: | 2 Investigative Sites in the U.S. |
| Name of Sponsor: | NIDEK CO., LTD. |
| Address of Sponsor: | 34-14 Meahama, Hiroishi-cho, Gamagori, Aichi, 443-0038, |
| | Japan |
| NCT Number: | NCT07152808 |
| Original Protocol | August 3, 2022 |
| (Version 1): | |
| Version 2 | May 16, 2023 |

## 2. STUDY PROTOCOL

This was a prospective clinical study to be conducted at two investigative sites located in the United States. The specific objective of the study was to assess the tonometer function and performance of the TONOREF III to the GAT. TONOREF III and GAT were used during study procedures. Investigators assessed IOP and remained masked to the results of the IOP measurement.

This was an open-label study, meaning all study staff and subjects were aware of which devices were being used. The GAT, and TONOREF III were used in accordance with this clinical protocol and Operator's Manual for each device.

Each subject was evaluated initially for suitability as a candidate for this study. Informed consent was obtained from each candidate prior to any study specific measurements not routinely performed,

including measurements with the investigational device. Subjects that were candidates for enrollment were asked their willingness to participate in this study and underwent the required screening for the confirmation of compliance with inclusion and exclusion criteria.



## 3. STATISTICAL ANALYSIS PLAN

**Analysis of Study Endpoints** 



The data analysis will include a comparison of the frequencies of all AEs, and ADEs (including subject complaints and corneal abrasions for the test device and reference tonometer).

The report of clinical agreement results will include the following presentation of results and analyses:

- a) Scatter plot of measured IOP values, with on the y-axis versus on the x-axis, using the same scale for the x and y axes.
- b) Similar to the Bland-Altman plot, the difference (minus minus versus results will be plotted with the mean difference and the 95% and 99% LOAs indicated.

Analysis of Safety Endpoints

The data analysis will include a comparison of the frequencies of all AEs and ADEs. AEs reported will be listed by subject and subject complaints and corneal abrasions for the test and reference devices will be specified.